CLINICAL TRIAL: NCT05045443
Title: Safety and Efficacy of Curcumin in Children With Acute Lymphoblastic Leukemia
Acronym: CurcumPedALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Soliman Elsayed Ebeid, MD, Professor of pediatrics Hematology Oncology and Bone Marrow Transplant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MD 134/2021
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: Curcumin; Ain Shams University; Egypt; Acute Lymphoblastic Leukemia; Children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Curcumin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Active Comparator): Tumeric curcumin 500 mg per oral capsule of Puritans Pride company supplement (composed of Tumeric (curcuma longa)root 450mg and Tumeric extract (curcuma longa )root 50mg ) standardized to contain 95%curcuminoids, it will given twice daily for 1 month starting at week 1 of maintenance phase of chemotherapy (Time 1) . It is preferably to be taken with meals but may be opened and prepared as a tea
  Interventions: Drug: Curcumin; Dietary Supplement: Standard of Care
- Standard of nutritional care (Placebo Comparator): Standard of nutritional support care
  Interventions: Dietary Supplement: Standard of Care

INTERVENTIONS:
Drug: Curcumin — Tumeric curcumin 500 mg per oral capsule of Puritans Pride company supplement
  Other Names: Tumeric curcumin
  Arms: Curcumin
Dietary Supplement: Standard of Care — As per institution protocol for Standard of nutritional Care

SUMMARY:
Assessment of of the biological effects of curcumin on microbiota in children with acute lymphoblastic leukemia

DETAILED DESCRIPTION:
Assessment of the safety of curcumin, which is the most active constituent of the ground rhizome of the Curcuma longa plant, in children with acute lymphoblastic leukemia patients (ALL) in maintenance phase of chemotherapy through the assessment of the any reported adverse event (AE). And assessment of the curcumin effect on health by eliminating intestinal microflora dysbiosis

ELIGIBILITY:
Inclusion Criteria:

Children aged from 1 year to 18 years Children with proven ALL diagnosed by bone marrow aspirate and immunephenotyping Patients in the maintenance phase week1

Exclusion Criteria:

Children with other maliganacies, Current use (past use of these medications is not an exclusion) of medications or over-the-counter treatments including to sulfasalazine, warfarin, clopidogrel, aspirin, antacids, botanical treatments (ginger, feverfew, yellow clover, Salix species, Populus species, Betula species, and Gaultheria species), essential fatty acids (flax oil and fish oil).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Determine the Safety of curcumin in pediatric patients with ALL. | 4 weeks
  Percentage of patients who developed adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Khairy, M.D, Study Chair — Faculty of Medicine Ain Shams University
Locations (1):
- Pediatric Hematology Oncology and BMT Unit, Faculty of Medicine Ain Shams University, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No